CLINICAL TRIAL: NCT03709563
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety and Efficacy of an Oral Nutraceutical Supplement With Standardized Botanicals in Males With Self-Perceived Thinning Hair and Loss
Brief Title: Oral Nutraceutical Supplement With Standardized Botanicals in Males With Self-Perceived Thinning Hair and Loss
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: DeNova Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HAIR 2018
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Hair Loss; Hair Thinning
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Nutraceutical Supplement (Active Comparator)
  Interventions: Dietary Supplement: Oral Nutraceutical Supplement
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oral Nutraceutical Supplement — Standardized Botanicals. Take 4 capsules by mouth daily with a meal
  Arms: Oral Nutraceutical Supplement
Dietary Supplement: Placebo — Placebo. Take 4 capsules by mouth daily with a meal
  Arms: Placebo

SUMMARY:
Hair loss study in men with self-perceived thinning hair and loss

ELIGIBILITY:
Inclusion Criteria:

1. Males between 21-45 years of age, inclusive
2. Have self-reported thinning or hair loss for more than 3 months prior to screening
3. Clinically confirmed to have hair loss or thinning by the investigator via physical exam, including subjects with male pattern hair loss with frontal and vertex patterns II, IIIv or IV using the Norwood Hamilton Hair Loss Scale (NHS).
4. In good general health, as determined by the Investigator
5. Willing and able to attend all study visits
6. Willing to maintain the same hair style as at the Screening Visit for the duration of the study.
7. Willing to use a mild non-medicated shampoo and conditioner for the duration of the study (medicated shampoo and conditioner refer to any prescription shampoo or conditioner as well as any over-the counter medicated shampoo or conditioner, such as those for treatment of dandruff or promoting hair growth)
8. Be willing and able to cooperate with the requirements of the study.
9. Voluntarily sign and date an informed consent agreement approved by the Institutional Review Board.
10. Be able to complete and understand the various rating instruments in English.

    -

Exclusion Criteria:

1. Clinical diagnosis of alopecia areata or scarring forms of alopecia
2. Scalp hair loss on the treatment area, due to disease, injury, or medical therapy
3. Current skin disease (e.g., psoriasis, atopic dermatitis, skin cancer, eczema, sun damage, seborrheic dermatitis), cuts and or abrasions on the scalp or condition (e.g., sunburn, tattoos) on the treatment area that, in the opinion of the Investigator, might put the subject at risk or interfere with the study conduct or evaluations.
4. History of surgical correction of hair loss on the scalp (i.e. Hair transplant).
5. Use of any products or devices purported to promote scalp hair growth (e.g., finasteride or minoxidil) within the 6 months prior to the Baseline Visit.
6. Use of anti-androgenic therapies (e.g., spironolactone, flutamide, cyproterone acetate, progesterone, and bicalutamide) within 3 months prior to the Baseline Visit.
7. History of burning, flaking, itching, and stinging of the scalp.
8. History of malignancy (except cutaneous squamous cell carcinoma and basal cell carcinoma) or currently undergoing chemotherapy or radiation treatments.
9. A known history of autoimmune thyroid disease, any other thyroid disorder/abnormality or other autoimmune disorders that in the opinion of the Investigator may interfere with the study treatment.
10. A known history of depression or bipolar disease or any other condition that may impact the subject's participation in the opinion of the investigator.
11. Recent utilization of low level lasers for hair growth.
12. Any condition that the Investigator thinks may put the Subject at risk or interfere with their participation in the study.
13. Known history or recent blood work indicating iron deficiency, bleeding disorders or platelet dysfunction syndrome as well as subjects receiving anticoagulant therapy or smokers with usage >20 cigarettes/day.
14. Use of any medications that are known to potentially cause hair loss or affect hair growth, as determined by the Investigator.

    -

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males only
Enrollment: 74 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Hair counts | Day 90, 180, 270, 360
  The change in vellus and terminal hair counts / average number of hairs (N/cm2) within 2 ROIs

SECONDARY OUTCOMES:
Shaft Thickness | Day 90, 180, 270, 360
Hair density | Day 90, 180, 270, 360

CONTACTS AND LOCATIONS:
Locations (1):
- DeNova Research, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No